CLINICAL TRIAL: NCT05934539
Title: A First-in-human, Multicenter, Open-label, Dose Escalation and Dose Expansion Phase 1 Study in Patients With Advanced Solid Tumors to Evaluate the Safety of Intravenously Administered ALG.APV-527
Brief Title: ALG.APV-527 First-in-human Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aptevo Therapeutics (Industry)
Collaborators: Alligator Bioscience AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALG.APV-527-101
Record Dates: First submitted 2023-02-26; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; 5T4

STUDY DESIGN:
Intervention Model Description: Escalating ALG.APV-527 doses with a starting dose of 0.1 mg/kg and projected 6 dose cohorts will be explored to determine the MTD and/or the RP2D. Part 1 consists of a 3 + 3 dose-escalation examination of ALG.APV-527 single agent therapy in adult patients with RECIST Version1.1-measurable advanced solid tumors. Part 2 consists of Dose Expansion using the RP2D, as determined during Dose Escalation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALG.APV-527 (Experimental): Part 1 Dose Escalation using ALG.APV-527 doses with a starting dose of 0.1 mg/kg and projected 6 dose cohorts will be explored to determine the MTD and/or the RP2D. Part 1 consists of a 3 + 3 dose-escalation examination of ALG.APV-527 single agent therapy in adult patients with RECIST Version1.1-measurable advanced solid tumors.
  Part 2 Dose Expansion with ALG.APV-527 based on RP2D determined during Dose Escalation.
  Interventions: Drug: ALG.APV-527

INTERVENTIONS:
Drug: ALG.APV-527 — ALG.APV-527 is a human bispecific antibody in the ADAPTIR™ format with a silenced immunoglobulin 1 (IgG1) Fc domain targeting the co-stimulatory receptor 4-1BB, expressed on immune cells such as CD8+ T cells and natural killer (NK) cells, and the tumor associated antigen 5T4. ALG.APV-527 is being co-developed by Alligator Bioscience AB (Lund, Sweden) and Aptevo Therapeutics Inc. (Seattle, WA, USA) as a cancer immunotherapy.
  Other Names: No other intervention names are planned for this study

SUMMARY:
A first-in-human, multicenter, open-label, dose escalation and dose expansion phase 1 study in patients with advanced solid tumors to evaluate the safety of intravenously administered ALG.APV-527 (Short title: ALG.APV-527 first-in-human study). Adult patients with advanced/metastatic solid tumors likely to express 5T4 antigen who have failed standard of care regimens for their cancer, have become refractory to standard treatment, or for whom no effective therapy exists based on investigator judgment may be enrolled in this study.

Part 1 (Dose Escalation): Approximately 36 evaluable patients planned to be enrolled.

Part 2 (Dose Expansion): Approximately 20 evaluable patients planned to be enrolled.

DETAILED DESCRIPTION:
This first-in-human study is an open-label, multicenter, Phase 1 study with the aim to assess safety and tolerability and preliminary anti-tumor activity of ALG.APV-527 administered intravenously to patients with advanced solid tumor malignancies. Patients will be required to provide tumor tissue biopsy material that has been obtained within 28 days prior to the first dose of study drug ALG.APV-527.

The trial has 2 parts, Part 1 (Dose Escalation) and Part 2 (Dose Expansion). The Escalation Phase (Part 1) is projected to occur in 6 patient cohorts of increasing dose levels and will explore the Maximum Tolerated Dose (MTD) and/or the RP2D. Part 1 consists of a 3 + 3 dose-escalation examination of ALG.APV-527 single agent therapy in adult patients with RECIST Version1.1-measurable advanced solid tumors.

The MTD is defined as the highest dose level that has 6 patients evaluable for DLT with no more than 1 of 6 with DLT.

Part 2 (Dose Expansion):

Part 2 consists of a single agent evaluation of the safety and clinical activity of ALG.APV-527 at its RP2D in up to 20 patients with advanced solid tumors. Part 2 will commence after all tested dose levels have been reviewed and a RP2D has been determined.

Primary Objectives:

Primary (Dose Escalation)

* To determine the safety, tolerability, MTD of ALG.APV-527 administered intravenously as single agent therapy
* To designate an IV dose level for the Dose Expansion Phase (RP2D) of ALG.APV-527 administered IV as single agent therapy for patients with advanced solid tumors. The RP2D can be different from the MTD.

Primary (Dose Expansion)

• To further evaluate the safety and tolerability of ALG.APV-527 when administered intravenously at the RP2D level as monotherapy in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Have provided signed informed consent form (ICF) for participation in the study.
* Have a diagnosis of advanced solid tumor malignancy (histologically or cytologically documented) that is metastatic or unresectable, have received standard of care therapy, and remaining therapeutic options are participation in a clinical study or non-curative therapy including best supportive care.
* Have one of the following tumors: non-small cell lung cancer (NSCLC), gastric/gastro-esophageal cancer, head and neck squamous cell carcinoma, renal cell cancer, ovarian cancer, breast cancer, malignant pleural mesothelioma, cervical cancer, colorectal cancer, urothelial carcinoma, endometrial cancer, pancreatic cancer, or prostate cancer.
* Must be ≥ 18 years of age.
* ECOG performance status 0-1.
* Has provided tumor tissue biopsy material that has been obtained within 28 days prior to the first dose of study drug with ALG.APV-527. Biopsy material may be provided as FFPE block or as pre-cut slides of 7 to 10 sequential tissue sections.
* Should have recovered from AEs due to prior anticancer medications to at least ≤Grade 1 by CTCAE version 5.0, except for alopecia, vitiligo, resolved atopy, and white blood cell count (see inclusion criterion #13).
* Must have at least 1 measurable lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST Version 1.1.
* Must have a life expectancy of ≥3 months.
* For women of childbearing potential and men with partners of childbearing potential, agreement to use a highly effective method of birth control for the duration of study treatment and for at least 9 months after the last dose of study treatment:

  * Combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal)
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable)
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomized partner
  * Sexual abstinence (defined as refraining from heterosexual intercourse during the entire study and for 9 months after the last dose of study treatment and must be the preferred and usual lifestyle of the patient)
* Females of childbearing potential must have a negative serum or urine pregnancy test.
* Must have adequate coagulation function at Screening as determined by:

  * PT international normalized ratio (INR) ≤ 1.5.
  * PTT ≤ 1.5 × ULN. Patients on full dose of oral anticoagulation must be on this dose for a minimum duration of 14 days before the first dose of study drug; if receiving warfarin, the patient must have an INR ≤ 3.0 and no active bleeding (i.e., no bleeding within 14 days prior to first dose of study drug); patients on low molecular weight heparin will be allowed.
* Must have adequate hematologic function at Screening as determined by:

  * White blood count cell (WBC) ≥ 2000/µL.
  * Absolute neutrophil count (ANC) ≥ 1500/µL (patient may not use G-CSF or GMCSF to achieve these WBC and ANC levels).
  * Platelet count ≥ 100 × 103/µL.
  * Hemoglobin (Hgb) ≥ 9.0 g/dL (may not transfuse or use erythropoietin to obtain this Hgb level; transfusions are allowed up to 2 weeks prior to C1D1).
* Must have adequate renal and hepatic function at Screening as determined by:

  * Adequate renal function (estimated glomerular filtration rate [eGFR] > 40 mL/min according to the Cockcroft-Gault formula).
  * Total bilirubin ≤ 1.5 × ULN (or ≤ 3.0 × ULN for patients with liver metastases or known Gilbert's syndrome).
  * AST and ALT ≤ 2.5 × ULN (≤ 5.0 × ULN in patients with documented liver metastasis).
  * Alkaline phosphatase ≤ 2.5 x ULN (≤ 5.0 × ULN in patients with documented liver or bone metastases)
* Must be able to attend study visits as required by the protocol.

Exclusion Criteria:

* Has received anti-cancer chemotherapy (including molecular-targeted drugs), radiotherapy (therapeutic or curative intent) or hormonal therapy within 14 days before the first dose of ALG.APV-527; however, the following are permitted:

  * Hormonal therapy with gonadotropin-releasing hormone (GnRH) agonists or antagonists for prostate cancer
  * Hormone-replacement therapy or oral contraceptives
  * Herbal therapy intended as anti-cancer ≥ 1 week prior to first dose of ALG.APV-527
  * Palliative radiotherapy for bone metastases within 2 weeks prior to first dose of ALG.APV-527
* Has received immunotherapy (e.g., CAR T-cell therapy, T-cell redirecting bispecific antibodies, mono-specific antibodies, vaccines or cytokines), or investigational agents within 28 days before the first dose of ALG.APV-527.
* Receives concurrent systemic (oral or IV) steroid therapy >10 mg methylprednisolone daily or its equivalent for an underlying, non-cancer condition. Concurrent corticosteroid therapy as anticancer drug (any dose) is considered exclusionary.
* Has had major surgery within the 4 weeks before the first dose of ALG.APV-527.
* History of, or known, central nervous system (CNS) disease involvement (e.g., glioblastoma [GBM]), carcinomatous meningitis, CNS metastases including spinal metastases with a risk of spinal cord compression (spinal metastases not associated with a risk of spinal cord compression are acceptable); CNS metastases that are treated and not progressing are acceptable.
* Has seizures requiring anticonvulsant treatment or has a history of a cerebrovascular accident or transient ischemic attack less than 6 months ago.
* Has uncontrolled or severe intercurrent medical condition or a significant history of renal, neurologic, psychiatric, pulmonary, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease that in the opinion of the investigator would adversely affect the patient's participation in this trial.
* Has interstitial lung disease or active, non-infectious pneumonitis.
* Has a history of autoimmune disease active or past including but not limited to inflammatory bowel disease, systemic lupus erythematosus (SLE), ankylosing spondylitis, scleroderma, or multiple sclerosis. Has any active immunologic disorder requiring immunosuppression with steroids >10mg methylprednisolone daily or its equivalent or other immunosuppressive agents (e.g., azathioprine, cyclosporine A) with the exception of patients with isolated vitiligo, resolved childhood asthma or atopic dermatitis, controlled hypoadrenalism or hypopituitarism, and euthyroid patients with a history of Grave's disease. Patients with controlled hyperthyroidism must be negative for thyroglobulin, thyroid peroxidase antibodies, and thyroid-stimulating immunoglobulin prior to study drug administration.
* Has a known hypersensitivity to a component of the protocol therapy, ALG.APV-527.
* Has a history of another primary cancer within the 5 years prior to enrollment except for the following: non-melanoma skin cancer, cervical carcinoma in situ, superficial bladder cancer, or other non-metastatic carcinoma that has been in complete remission without treatment for more than 5 years.
* Has abnormal electrocardiograms (ECGs) that are clinically significant, such as QT prolongation (corrected QT interval [QTcF] > 470 msec).
* In the opinion of the treating Investigator, has any concurrent conditions that could pose an undue medical hazard or interfere with the interpretation of the study results; these conditions include, but are not limited to ongoing or active infection, clinically significant non-healing or healing wounds, concurrent congestive heart failure (New York Heart Association Functional Classification Class II, III or IV), concurrent unstable angina, concurrent cardiac arrhythmia requiring treatment (excluding asymptomatic atrial fibrillation), recent (within the prior 12 months) myocardial infarction, acute coronary syndrome or stroke within the previous 12 months, significant valvular disease, cardiomegaly, ventricular hypertrophy, or cardiomyopathy, significant pulmonary disease (shortness of breath at rest or on mild exertion), for example, because of concurrent severe obstructive pulmonary disease, concurrent hypertension requiring more than 2 medications for adequate control, or diabetes mellitus with more than 2 episodes of ketoacidosis in the prior 12 months.
* Has an ejection fraction (EF) of 50% or less based on a multi-gated acquisition (MUGA) scan or echocardiogram (ECHO).
* Patient has any active, uncontrolled, or suspected infection at the time of signing ICF or within 3 days prior to treatment start.
* Has the presence of a known active acute or chronic infection (viral, bacterial, systemic fungal) including human immunodeficiency virus (HIV) as determined by enzyme-linked immunosorbent assay (ELISA) and confirmed by Western blot; and hepatitis B virus (HBV) and hepatitis C virus (HCV) as determined by hepatitis B surface antigen (HBsAg) and hepatitis C serology (prophylactic therapy according to institutional protocols is acceptable).
* Has a cognitive, psychological, or psychosocial impediment that would impair the ability of the patient to receive therapy according to the protocol or adversely affect the ability of the patient to comply with the informed consent process, protocol, or protocol-required visits and procedures.
* Pregnant or breastfeeding.
* Have been exposed to live attenuated vaccine within 4 weeks prior to first dose of ALG.APV-527.
* Participation or plans to participate in another interventional clinical study while taking part in this protocol; participation in an observational study is acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) | 28 days for Q2W
  Number of participants with DLTs during the 28 days following the first administration of Q2W ALG.APV 527 or during the 42 days following Q3W ALG.APV 527
Overall Response Rate | Through completion of Expansion Phase. Approximately 24 months.
  The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence based on the response evaluation criteria in solid tumors (RECIST), v1.1

SECONDARY OUTCOMES:
Pharmacokinetic measure- Peak Plasma Concentration (Cmax) | Through completion of both Dose Escalation and Dose Expansion ( Approx 42 months)
  Pharmacokinetic samples will be collected at predefined timepoints to determine Cmax.
Pharmacokinetic measure- Area under the plasma concentration versus time curve (AUC) | Through completion of both Dose Escalation and Dose Expansion ( Approx 42 months)
  Pharmacokinetic samples will be collected at predefined timepoints to determine AUC.

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Oncology Associates Of The Treasure Coast, Port Saint Lucie, Florida, United States